CLINICAL TRIAL: NCT02414386
Title: Serum Vitamin D Levels in Multi-organ Failure Critically Ill Patients Undergoing Regional Citrate Anticoagulation Continuous Renal Replacement Therapies - Prospective Observational Case-control Study
Brief Title: Serum Vitamin D Levels in Critically Ill Patients Undergoing Regional Citrate Anticoagulation CRRT
Acronym: VitDcrrt
Status: Completed | Type: Observational
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Czarnik, MD PhD, Tomasz Czarnik, MD PhD, Uniwersytecki Szpital Kliniczny w Opolu
Other Study IDs: VitaminDcitrateCRRT
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Multi Organ Failure; Acute Kidney Injury
Keywords: Vitamin D; Continuous Renal Replacement Therapy; Multi Organ Failure; Acute Kidney Injury; Critical Care; Citrate anticoagulation
MeSH Terms: conditions — Multiple Organ Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples taken from the arterial catheter every 12 hours to obtain vitamin D, parathormon, calcium, magnesium, phosphate, globulin, albumin plasma levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute Kidney Injury - CRRT: Multi-organ failure with acute kidney injury critically ill patients admitted to the critical care unit undergoing regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF). Multi-organ failure is defined as a respiratory, circulatory and renal failure. Biospecimen retention to measure vitamin D, parathormone, calcium, magnesium, phosphate, globulin, albumin plasma levels.
  Interventions: Other: biospecimen retention
- Control: Multi-organ failure non acute kidney injury critically ill patients admitted to the critical care unit. Multi-organ failure is defined as a respiratory and circulatory failure. Biospecimen retention to measure vitamin D, parathormone, calcium, magnesium, phosphate, globulin, albumin plasma levels.
  Interventions: Other: biospecimen retention

INTERVENTIONS:
Other: biospecimen retention — biospecimen retention to measure vitamin D, parathormone, calcium, magnesium, phosphate, globulin, albumin plasma levels

SUMMARY:
Several studies point at a potential relationship between vitamin D deficiency and worse outcome in critically ill patients admitted to the intensive care unit. It is linked with the lack of vitamin D pleiotropic effects in the state of hypovitaminosis D. The pleiotropism of vitamin D is dependent on a specific feature of vitamin D receptor (VDR) namely polymorphism and its universal existence in the human body. Vitamin D pleiotropism is linked with cancer cells inhibition, a modulation of the immune system, an influence on cardiovascular system and neuroprotection.

In 35-65% critically ill patients hospitalized in the intensive care unit the acute kidney injury (AKI) is diagnosed. Acute kidney injury increases significantly the probability of death. The standard therapy of a severe AKI in many intensive care units is the regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF). The specificity of the regional citrate anticoagulation by means of precise ionized calcium and citrate dosing evokes questions regarding its influence on vitamin D and entire calcium-phosphate metabolism in the state of a severe AKI treated with regional citrate anticoagulation continuous renal replacement therapy.

The intention of that trial is to measure vitamin D plasma levels and other parameters (parathormone, ionized and total calcium, magnesium, phosphate, albumin, globulin) linked with calcium-phosphate metabolism in the human body. We would like to assess potential relationships between the regional citrate anticoagulation continuous renal replacement therapy and these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory, circulatory failure and acute kidney injury mechanically ventilated critically ill patients admitted to the critical care unit undergoing regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF)

Exclusion Criteria:

* age less than 18 years
* acute liver failure
* hypercalcemia at admission (total calcium plasma level > 10.6 mg/dL; total ionized calcium plasma level > 1.35 mmol/L)
* parathyroid glands disease at admission
* serum vitamin D level < 10 ng/ml at admission
* end stage renal disease at admission
* lack of relatives consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Kidney Injury - CRRT group: Multi-organ failure with acute kidney injury critically ill patients admitted to the critical care unit undergoing regional citrate anticoagulation continuous renal replacement therapy by means of continuous veno-venous hemodiafiltration (CVVHDF). Multi-organ failure is defined as a respiratory, circulatory and renal failure.
  Control group: Multi-organ failure non acute kidney injury critically ill patients admitted to the critical care unit. Multi-organ failure is defined as a respiratory and circulatory failure.
  All patients: machanically ventilated.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
The relationship between vitamin D plasma levels and regional citrate CRRT | 96 hours
  The first vitamin D plasma level measurement at admission, before the start of CRRT (the zero point) Next vitamin D plasma level measurements every 12 hours. Minimal number of measurements - 6, maximal - 8.

SECONDARY OUTCOMES:
The relationship between other parameters of calcium-phosphate metabolism and regional citrate CRRT | 96 hours
  The first parathormone, total and ionized calcium, phosphate, magnesium plasma levels measurement at admission, before the start of CRRT (the zero point) Next measurements every 12 hours. Minimal number of measurements - 4, maximal - 8.
  The albumin and globulin plasma levels measurements at admission and at the last measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Czarnik, MD PhD, Principal Investigator — Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu
Locations (2):
- Poland (2):
  - Department of Endocrinology, Szpital Wojewodzki w Opolu, Opole, Silesian Voivodeship
  - Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Silesian Voivodeship

REFERENCES:
- [Result] Czarnik T, Czarnik A, Gawda R, Piwoda M, Marszalski M, Czuczwar M. Vitamin D serum levels in multiorgan failure critically ill patients undergoing continuous renal replacement therapies. Anaesthesiol Intensive Ther. 2020;52(5):359-365. doi: 10.5114/ait.2020.101008. PMID 33242935